CLINICAL TRIAL: NCT05916209
Title: Pericapsular Nerve Group (PENG) Block and Lateral Femoral Cutaneous Nerve (LFCN) Block Versus Fascia Iliaca (FIC) Block for Multimodal Analgesia After Total Hip Replacement Surgery: a Retrospective Analysis
Brief Title: PENG and LFCN Block Versus FIC Block for Multimodal Analgesia After Total Hip Replacement Surgery: a Retrospective Analysis
Acronym: PENG+LFCN-FICB
Status: Completed | Type: Observational
Sponsor: Ospedale Edoardo Bassini (Other)
Responsible Party: Principal Investigator, Francesco Vetrone, Medical Doctor - Principal Investigator, Ospedale Edoardo Bassini
Other Study IDs: 044.677
Record Dates: First submitted 2023-05-19; First posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Regional Anesthesia Morbidity; Arthropathy of Hip; Hip Arthropathy
Keywords: total hip replacement surgery; primary hip arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PENG + LFCN Block: group in which PENG + LFCN Block was performed
  Interventions: Procedure: Peripheral nerve blocks
- FIC Block: group in which FIC Block was performed
  Interventions: Procedure: Peripheral nerve blocks

INTERVENTIONS:
Procedure: Peripheral nerve blocks — Peripheral nerve blocks provide intense, site-specific analgesia administring local anesthetics near the nerves.

SUMMARY:
Background: Optimal pain control with limited muscle weakness is paramount for a swift initiation of physical therapy and ambulation. Fascia iliaca compartment block (FICB) has been recommended since it offers the best pain control with low risk of motor block. Pericapsular nerve group block (PENG) with lateral femoral cutaneous nerve (LFCN) block has been proposed as an effective alternative to FICB that offers similar pain control with a considerably lower risk of motor block. This study aimed to compare the afore mentioned blocks and determine which one yielded the lowest NRS score.

DETAILED DESCRIPTION:
This single-center, retrospective investigation was conducted at ASST Nord Milano Bassini hospital. The study was approved by the ethics committee "Comitato Etico Milano Area 3". The main outcome of the study was the comparison of postoperative pain at 6, 12 and 24 hours, expressed as NRS (numeric rating scale), between PENG and LCFN . Secondary outcomes included total opioid consumption expressed as milligrams of morphine equivalents (MME), time to first opioid request, time to first postoperative ambulation.

ELIGIBILITY:
Inclusion Criteria:

* elective total hip replacement surgery for non-traumatic hip disease, age >18 years, complete clinical chart included the type of peripheral nerve block performed, signed consent form for spinal anesthesia and peripheral nerve block.

Exclusion Criteria:

* incomplete chart, a peripheral nerve block other than PENG or FIC block was performed

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary hip replacement surgery
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
pain control | 6 hours after surgery
  pain assessment with Numeric Rating Scale (NRS): a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable"
pain control | 12 hours after surgery
  pain assessment with Numeric Rating Scale (NRS): a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable"
pain control | 24 hours after surgery
  pain assessment with Numeric Rating Scale (NRS): a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable"

SECONDARY OUTCOMES:
MME of PRN opioid doses | 6 hours after surgery
  we studied the effect of Regional anesthesia on opioid-sparing
MME of PRN opioid doses | 12 hours after surgery
  we studied the effect of Regional anesthesia on opioid-sparing
Morphine Milligram Equivalents (MME) of "pro re nata" (PRN) opioid doses | 24 hours after surgery
  we studied the effect of Regional anesthesia on opioid-sparing

OTHER OUTCOMES:
time to first opioid request | From date of surgery until up to 3 days after
  we studied the effect of Regional anesthesia on opioid-sparing
time to first postoperative ambulation | From date of surgery until up to 100 days after
  we studied the effect or Regional anesthesia on residual paralysis

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Edoardo Bassini, Cinisello Balsamo, Milano, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Memtsoudis SG, Cozowicz C, Bekeris J, Bekere D, Liu J, Soffin EM, Mariano ER, Johnson RL, Hargett MJ, Lee BH, Wendel P, Brouillette M, Go G, Kim SJ, Baaklini L, Wetmore D, Hong G, Goto R, Jivanelli B, Argyra E, Barrington MJ, Borgeat A, De Andres J, Elkassabany NM, Gautier PE, Gerner P, Gonzalez Della Valle A, Goytizolo E, Kessler P, Kopp SL, Lavand'Homme P, MacLean CH, Mantilla CB, MacIsaac D, McLawhorn A, Neal JM, Parks M, Parvizi J, Pichler L, Poeran J, Poultsides LA, Sites BD, Stundner O, Sun EC, Viscusi ER, Votta-Velis EG, Wu CL, Ya Deau JT, Sharrock NE. Anaesthetic care of patients undergoing primary hip and knee arthroplasty: consensus recommendations from the International Consensus on Anaesthesia-Related Outcomes after Surgery group (ICAROS) based on a systematic review and meta-analysis. Br J Anaesth. 2019 Sep;123(3):269-287. doi: 10.1016/j.bja.2019.05.042. Epub 2019 Jul 24. PMID 31351590
- [Background] Anger M, Valovska T, Beloeil H, Lirk P, Joshi GP, Van de Velde M, Raeder J; PROSPECT Working Group* and the European Society of Regional Anaesthesia and Pain Therapy. PROSPECT guideline for total hip arthroplasty: a systematic review and procedure-specific postoperative pain management recommendations. Anaesthesia. 2021 Aug;76(8):1082-1097. doi: 10.1111/anae.15498. Epub 2021 May 20. PMID 34015859
- [Background] Gan TJ. Poorly controlled postoperative pain: prevalence, consequences, and prevention. J Pain Res. 2017 Sep 25;10:2287-2298. doi: 10.2147/JPR.S144066. eCollection 2017. PMID 29026331
- [Background] Joshi GP, Kehlet H. Postoperative pain management in the era of ERAS: An overview. Best Pract Res Clin Anaesthesiol. 2019 Sep;33(3):259-267. doi: 10.1016/j.bpa.2019.07.016. Epub 2019 Jul 25. PMID 31785712
- [Background] Shelton C, White S. Anaesthesia for hip fracture repair. BJA Educ. 2020 May;20(5):142-149. doi: 10.1016/j.bjae.2020.02.003. Epub 2020 Mar 23. No abstract available. PMID 33456943
- [Background] Chuan A, Zhao L, Tillekeratne N, Alani S, Middleton PM, Harris IA, McEvoy L, Ni Chroinin D. The effect of a multidisciplinary care bundle on the incidence of delirium after hip fracture surgery: a quality improvement study. Anaesthesia. 2020 Jan;75(1):63-71. doi: 10.1111/anae.14840. Epub 2019 Sep 23. PMID 31549413
- [Background] Peters CL, Shirley B, Erickson J. The effect of a new multimodal perioperative anesthetic regimen on postoperative pain, side effects, rehabilitation, and length of hospital stay after total joint arthroplasty. J Arthroplasty. 2006 Sep;21(6 Suppl 2):132-8. doi: 10.1016/j.arth.2006.04.017. PMID 16950075
- [Background] Costa-Martins I, Carreteiro J, Santos A, Costa-Martins M, Artilheiro V, Duque S, Campos L, Chedas M. Post-operative delirium in older hip fracture patients: a new onset or was it already there? Eur Geriatr Med. 2021 Aug;12(4):777-785. doi: 10.1007/s41999-021-00456-w. Epub 2021 Feb 11. PMID 33569717
- [Background] Steiner LA. Postoperative delirium. Part 1: pathophysiology and risk factors. Eur J Anaesthesiol. 2011 Sep;28(9):628-36. doi: 10.1097/EJA.0b013e328349b7f5. PMID 21785356
- [Background] Tsinaslanidis G, Tsinaslanidis P, Mahajan RH. Perioperative Pain Management in Patients Undergoing Total Hip Arthroplasty: Where Do We Currently Stand? Cureus. 2020 Jul 7;12(7):e9049. doi: 10.7759/cureus.9049. PMID 32782868
- [Background] Duque M, Schnetz MP, Yates AJ Jr, Monahan A, Whitehurst S, Mahajan A, Kaynar AM. Impact of Neuraxial Versus General Anesthesia on Discharge Destination in Patients Undergoing Primary Total Hip and Total Knee Replacement. Anesth Analg. 2021 Dec 1;133(6):1379-1386. doi: 10.1213/ANE.0000000000005156. PMID 34784324
- [Background] Johnson RL, Kopp SL, Burkle CM, Duncan CM, Jacob AK, Erwin PJ, Murad MH, Mantilla CB. Neuraxial vs general anaesthesia for total hip and total knee arthroplasty: a systematic review of comparative-effectiveness research. Br J Anaesth. 2016 Feb;116(2):163-76. doi: 10.1093/bja/aev455. PMID 26787787
- [Background] O'Reilly N, Desmet M, Kearns R. Fascia iliaca compartment block. BJA Educ. 2019 Jun;19(6):191-197. doi: 10.1016/j.bjae.2019.03.001. Epub 2019 Apr 24. No abstract available. PMID 33456890
- [Background] Zhang XY, Ma JB. The efficacy of fascia iliaca compartment block for pain control after total hip arthroplasty: a meta-analysis. J Orthop Surg Res. 2019 Jan 25;14(1):33. doi: 10.1186/s13018-018-1053-1. PMID 30683117
- [Background] Gao Y, Tan H, Sun R, Zhu J. Fascia iliaca compartment block reduces pain and opioid consumption after total hip arthroplasty: A systematic review and meta-analysis. Int J Surg. 2019 May;65:70-79. doi: 10.1016/j.ijsu.2019.03.014. Epub 2019 Mar 25. PMID 30922995
- [Background] Jones MR, Novitch MB, Hall OM, Bourgeois AP, Jeha GM, Kaye RJ, Orhurhu V, Orhurhu MS, Eng M, Cornett EM, Kaye AD. Fascia iliaca block, history, technique, and efficacy in clinical practice. Best Pract Res Clin Anaesthesiol. 2019 Dec;33(4):407-413. doi: 10.1016/j.bpa.2019.07.011. Epub 2019 Jul 26. PMID 31791559
- [Background] Gasanova I, Alexander JC, Estrera K, Wells J, Sunna M, Minhajuddin A, Joshi GP. Ultrasound-guided suprainguinal fascia iliaca compartment block versus periarticular infiltration for pain management after total hip arthroplasty: a randomized controlled trial. Reg Anesth Pain Med. 2019 Feb;44(2):206-211. doi: 10.1136/rapm-2018-000016. PMID 30700615
- [Background] Giron-Arango L, Peng PWH, Chin KJ, Brull R, Perlas A. Pericapsular Nerve Group (PENG) Block for Hip Fracture. Reg Anesth Pain Med. 2018 Nov;43(8):859-863. doi: 10.1097/AAP.0000000000000847. PMID 30063657
- [Background] Pascarella G, Costa F, Del Buono R, Pulitano R, Strumia A, Piliego C, De Quattro E, Cataldo R, Agro FE, Carassiti M; collaborators. Impact of the pericapsular nerve group (PENG) block on postoperative analgesia and functional recovery following total hip arthroplasty: a randomised, observer-masked, controlled trial. Anaesthesia. 2021 Nov;76(11):1492-1498. doi: 10.1111/anae.15536. Epub 2021 Jul 1. PMID 34196965
- [Background] Kukreja P, Avila A, Northern T, Dangle J, Kolli S, Kalagara H. A Retrospective Case Series of Pericapsular Nerve Group (PENG) Block for Primary Versus Revision Total Hip Arthroplasty Analgesia. Cureus. 2020 May 19;12(5):e8200. doi: 10.7759/cureus.8200. PMID 32572357
- [Background] Fernicola, Jacob Tannehill I, Tucker CJ, Robert Volk W, Dickens JF. The Pericapsular Nerve Group Block for Perioperative Pain Management for Hip Arthroscopy. Arthrosc Tech. 2021 Jul 22;10(7):e1799-e1803. doi: 10.1016/j.eats.2021.03.029. eCollection 2021 Jul. PMID 34336578
- [Background] Aliste J, Layera S, Bravo D, Jara A, Munoz G, Barrientos C, Wulf R, Branez J, Finlayson RJ, Tran Q. Randomized comparison between pericapsular nerve group (PENG) block and suprainguinal fascia iliaca block for total hip arthroplasty. Reg Anesth Pain Med. 2021 Oct;46(10):874-878. doi: 10.1136/rapm-2021-102997. Epub 2021 Jul 20. PMID 34290085
- [Background] Remily EA, Hochstein SR, Wilkie WA, Mohamed NS, Thompson JV, Kluk MW, Nace J, Delanois RE. The pericapsular nerve group block: a step towards outpatient total hip arthroplasty? Hip Int. 2022 May;32(3):318-325. doi: 10.1177/1120700020978211. Epub 2020 Dec 3. PMID 33269617
- [Background] Nielsen TD, Moriggl B, Barckman J, Kolsen-Petersen JA, Soballe K, Borglum J, Bendtsen TF. The Lateral Femoral Cutaneous Nerve: Description of the Sensory Territory and a Novel Ultrasound-Guided Nerve Block Technique. Reg Anesth Pain Med. 2018 May;43(4):357-366. doi: 10.1097/AAP.0000000000000737. PMID 29381568
- [Background] da Costa AO, Izolani GV, Monteiro de Souza IF, Martins Santiago BV. Continuous pericapsular nerve group (PENG) block through an elastomeric infusion system, associated with the lateral cutaneous nerve block of the thigh for total hip arthroplasty. BMJ Case Rep. 2022 Mar 29;15(3):e246833. doi: 10.1136/bcr-2021-246833. PMID 35351743
- [Background] Gurbuz H, Okmen K, Gultekin A. Postoperative pain management in patients with coxarthrosis undergoing total hip arthroplasty: PENG block combined with LFCN block or wound infiltration? Minerva Anestesiol. 2021 Oct;87(10):1154-1155. doi: 10.23736/S0375-9393.21.15757-8. Epub 2021 May 13. No abstract available. PMID 33982993
- [Background] Thallaj A. Combined PENG and LFCN blocks for postoperative analgesia in hip surgery-A case report. Saudi J Anaesth. 2019 Oct-Dec;13(4):381-383. doi: 10.4103/sja.SJA_299_19. PMID 31572090
- [Background] Vilhelmsen F, Nersesjan M, Andersen JH, Danker JK, Broeng L, Hagi-Pedersen D, Mathiesen O, Thybo KH. Lateral femoral cutaneous nerve block with different volumes of Ropivacaine: a randomized trial in healthy volunteers. BMC Anesthesiol. 2019 Aug 28;19(1):165. doi: 10.1186/s12871-019-0833-4. PMID 31455249
- [Background] Ying H, Chen L, Yin D, Ye Y, Chen J. Efficacy of pericapsular nerve group block vs. fascia iliaca compartment block for Hip surgeries: A systematic review and meta-analysis. Front Surg. 2023 Feb 10;10:1054403. doi: 10.3389/fsurg.2023.1054403. eCollection 2023. PMID 36843984
- [Background] Dowell D, Ragan KR, Jones CM, Baldwin GT, Chou R. CDC Clinical Practice Guideline for Prescribing Opioids for Pain - United States, 2022. MMWR Recomm Rep. 2022 Nov 4;71(3):1-95. doi: 10.15585/mmwr.rr7103a1. PMID 36327391
- [Background] Kaye AD, Urman RD, Cornett EM, Hart BM, Chami A, Gayle JA, Fox CJ. Enhanced recovery pathways in orthopedic surgery. J Anaesthesiol Clin Pharmacol. 2019 Apr;35(Suppl 1):S35-S39. doi: 10.4103/joacp.JOACP_35_18. PMID 31142957
- [Background] Del Buono R, Padua E, Pascarella G, Costa F, Tognu A, Terranova G, Greco F, Fajardo Perez M, Barbara E. Pericapsular nerve group block: an overview. Minerva Anestesiol. 2021 Apr;87(4):458-466. doi: 10.23736/S0375-9393.20.14798-9. Epub 2021 Jan 12. PMID 33432791
- [Background] Sercia QP, Bergeron JJ, Pelet S, Belzile EL. Continuous vs. single-shot adductor canal block for pain management following primary total knee arthroplasty: A systematic review and meta-analysis of randomized controlled trials. Orthop Traumatol Surg Res. 2022 Dec;108(8):103290. doi: 10.1016/j.otsr.2022.103290. Epub 2022 Apr 22. PMID 35470114
- [Background] Jenstrup MT, Jaeger P, Lund J, Fomsgaard JS, Bache S, Mathiesen O, Larsen TK, Dahl JB. Effects of adductor-canal-blockade on pain and ambulation after total knee arthroplasty: a randomized study. Acta Anaesthesiol Scand. 2012 Mar;56(3):357-64. doi: 10.1111/j.1399-6576.2011.02621.x. Epub 2012 Jan 4. PMID 22221014
- [Background] Gallagher RM, Polomano RC, Giordano NA, Farrar JT, Guo W, Taylor L, Oslin D, Goff BJ, Buckenmaier CC. Prospective cohort study examining the use of regional anesthesia for early pain management after combat-related extremity injury. Reg Anesth Pain Med. 2019 Sep 27:rapm-2019-100773. doi: 10.1136/rapm-2019-100773. Online ahead of print. PMID 31563880
- [Background] Farag A, Hendi NI, Diab RA. Does pericapsular nerve group block have limited analgesia at the initial post-operative period? Systematic review and meta-analysis. J Anesth. 2023 Feb;37(1):138-153. doi: 10.1007/s00540-022-03129-5. Epub 2022 Nov 7. PMID 36342537
- [Background] Kukreja P, Uppal V, Kofskey AM, Feinstein J, Northern T, Davis C, Morgan CJ, Kalagara H. Quality of recovery after pericapsular nerve group (PENG) block for primary total hip arthroplasty under spinal anaesthesia: a randomised controlled observer-blinded trial. Br J Anaesth. 2023 Jun;130(6):773-779. doi: 10.1016/j.bja.2023.02.017. Epub 2023 Mar 22. PMID 36964012
- [Background] Valoriani J, Conti D, Gianesello L, Pavoni V. Combined pericapsular nerve group and lateral femoral cutaneous nerve blocks for hip fracture in a polytraumatized patient-A case report. Saudi J Anaesth. 2022 Apr-Jun;16(2):211-213. doi: 10.4103/sja.sja_625_21. Epub 2022 Mar 17. PMID 35431737
- [Background] Roy R, Agarwal G, Pradhan C, Kuanar D. Total postoperative analgesia for hip surgeries, PENG block with LFCN block. Reg Anesth Pain Med. 2019 Mar 28:rapm-2019-100454. doi: 10.1136/rapm-2019-100454. Online ahead of print. No abstract available. PMID 30923252

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-27): https://cdn.clinicaltrials.gov/large-docs/09/NCT05916209/Prot_SAP_000.pdf